CLINICAL TRIAL: NCT01484145
Title: An Unblinded Clinical Trial to Evaluate the Deposition of Terbinafine in the Nail Bed After Iontophoretic Application of ETS Terbinafine Gel in Subjects With Distal Subungual Onychomycosis in the Great Toenail
Brief Title: Deposition of Terbinafine After Iontophoretic Application of ETS Terbinafine Gel in Subjects With Distal Subungual Onychomycosis in the Great Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-10
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Nail fungus; Tinea Unguium
MeSH Terms: conditions — Onychomycosis | interventions — Terbinafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 6 mA.min, 20 mins (Active Comparator)
  Interventions: Drug: Terbinafine HCl
- 6 mA/min, 20 mins, clamping (Experimental)
  Interventions: Drug: Terbinafine HCl
- 6 mA/min, 20 mins, debridement, clamping (Experimental)
  Interventions: Drug: Terbinafine HCl
- 15 mA/min, 30 mins, clamping (Experimental)
  Interventions: Drug: Terbinafine HCl
- 15 mA/min, 50 mins, debridement, clamping (Experimental)
  Interventions: Drug: Terbinafine HCl

INTERVENTIONS:
Drug: Terbinafine HCl — 4% w/w terbinafine HCL gel, single dose,

SUMMARY:
The purpose of this study is to determine how much terbinafine is delivered to the nail bed after treatment with a number of modifications to a previously studied method for iontophoretic delivery of terbinafine gel. Iontophoretic delivery involves the use of a small electric charge to deliver drug across skin and nails.

ELIGIBILITY:
Inclusion Criteria:

* Positive KOH
* 25-75% involvement of the visible nail.
* Nail plate must be < 3 mm thick.
* Must have signed informed consent.
* Must agree to avoid any type of pedicure or application of any nail polish product or nail cosmetic to the toenails after the screening visit until Day 28.
* Female subjects of childbearing potential must agree to take measures to avoid pregnancy until the day after Day 28
* Must agree to avoid the use of oral antifungals or topical terbinafine anywhere on the body until the day after Day 28. Topical antifungals other than terbinafine can be used on the body other than the feet after Day 0.

Exclusion Criteria:

* Presence of proximal subungual onychomycosis or white superficial onychomycosis
* Fungal involvement of a majority of the lunula
* Subjects with psoriasis, eczema, or other abnormalities that could result in a clinically abnormal nail
* Presence of dermatophytoma or onychomycotic spikes or exclusively lateral groove involvement
* Traumatized or dystrophic target great toenail.
* Known diabetics
* Subjects with peripheral vascular disease
* Subjects who are immunosuppressed (chronic corticosteroid therapy, solid organ or bone marrow transplantation, cytotoxic chemotherapy within the previous 12 months (or planned within the next 12 months), or HIV infection.
* Use of systemic corticosteroids within 30 days preceding Day 0
* Use of topical antifungals on the feet in the preceding 30 days of Day 0 through Day 28
* Use of topical terbinafine in the 30 days prior to treatment through Day 28
* Use of systemic antifungals in the preceding 120 days of Day 0 through Day 28
* Use of any investigational drug(s) within 30 days (120 days for systemic antifungals) preceding Day 0 through Day 28
* Has previously participated in this study
* Is pregnant or is a nursing mother
* Women of of child bearing potential who are not using an adequate form of contraception (or abstinence)
* Subjects with pacemakers/automatic implantable cardioverter/defibrillators
* Subjects with an implantable electronic device.
* Subjects with a bleeding disorder or who are using warfarin or any other blood coagulation modulator including aspirin in the 14 days prior to treatment through Day 28

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Level of terbinafine in the nail bed (ng/mg) | Day 28
Plasma terbinafine levels (ng/ml) | Day 28

SECONDARY OUTCOMES:
Number of treatment emergent adverse events (AEs)& Serious Adverse Events (SAEs) | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research, San Antonio, Texas, United States